CLINICAL TRIAL: NCT00718146
Title: Immunogenicity and Safety of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2008-2009 Formulation (Intramuscular Route)
Brief Title: Immunogenicity and Safety of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2008-2009 Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRT83
Record Dates: First submitted 2008-05-07; First posted 2008-07-18 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviridae Infections; Orthomyxoviruses; Split-virion influenza vaccine
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Age 16 to 60 years
  Interventions: Biological: Split virion, inactivated Influenza vaccine
- Group 2 (Experimental): Age over 60 years
  Interventions: Biological: Split virion, inactivated Influenza vaccine

INTERVENTIONS:
Biological: Split virion, inactivated Influenza vaccine — 0.5 mL, Intramuscular (IM)
  Arms: Group 1
Biological: Split virion, inactivated Influenza vaccine — 0.5 mL, Intramuscular (IM)
  Arms: Group 2

SUMMARY:
This study is for a new marketing authorization application for the seasonal vaccine strains in compliance with the Note for Guidance (NfG) on harmonization requirements for influenza vaccine from the Committee for Human Medicinal Products (CHMP)

Objectives:

* To evaluate the compliance, in terms of immunogenicity, of the inactivated, split-virion influenza vaccine NH 2008-2009 formulation with the requirements of the CHMP NfG CPMP/BWP/214/96.
* To describe the safety of the inactivated, split-virion influenza vaccine, NH 2008-2009 formulation.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 60 years or 61 years and older on the day of inclusion
* Provision of a signed informed consent
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential: avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 21 days after vaccination

Exclusion Criteria :

* For a woman of child-bearing potential, known pregnancy or positive urine pregnancy test at visit 01
* Febrile illness (temperature ≥ 37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to egg proteins, chick proteins, neomycin, formaldehyde and octoxinol 9, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 3 weeks following the trial vaccination
* Previous vaccination against influenza in the previous 6 months
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen or Hepatitis C seropositivity
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of Influenza vaccine (split virion, inactivated). | 21 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (2):
- United Kingdom (2):
  - Edinburgh
  - London

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com